CLINICAL TRIAL: NCT03693833
Title: CBD Treatment in Hand Osteoarthritis and Psoriatic Arthritis. A Randomized, Double-blind Placebo Controlled Study
Brief Title: CBD Treatment in Hand Osteoarthritis and Psoriatic Arthritis.
Acronym: NordCAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Jonathan Vela, Jonathan Vela MD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NordCAN
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Psoriatic Arthritis; Hand Osteoarthritis
Keywords: Cannabidiol; Cannabis; Osteoarthritis; Psoriatic arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Marijuana Abuse; Osteoarthritis | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 10mg Cannabidiol (CBD) tablets once daily for the first two weeks increasing to twice daily for week 3 and 4 if adequate analgesic effect is not attained at week 5 then the dose can be increased to 10mg thrice daily from week 5 and onward.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): 10mg Placebo Oral tablets once daily for the first two weeks increasing to twice daily for week 3 and 4 if adequate analgesic effect is not attained at week 5 then the dose can be increased to 10mg thrice daily from week 5 and onward.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol (CBD) tablets of 10mg each
  Other Names: CBD
  Arms: Intervention
Drug: Placebo Oral Tablet — Oral Placebo tablets of 10mg each
  Other Names: Oral Placebo
  Arms: Placebo

SUMMARY:
A randomized, placebo-controlled trial with blinded outcome assessments will be conducted to evaluate the efficacy and safety of CBD in patients with Hand-OA and PsA during a 12-week treatment period.

DETAILED DESCRIPTION:
A randomized, placebo-controlled trial with blinded outcome assessments will be conducted to evaluate the efficacy and safety of CBD in patients with Hand-OA and PsA during a 12-week treatment period.

Aim: To assess the effect of CBD on visual analogue scale pain measurements at 12 weeks compared with placebo.

Patients and controls: Patients with Hand-OA or PsA and VASpain during the last 24hours of 30mm or more.

Primary outcome: Changes in VAS pain during the last 24 hours from baseline to 12 weeks. Measured with a 100mm VAS from the most symptomatic hand (Hand-OA) or joint (PsA).

Safety outcomes

1. Percentage of patients experiencing adverse events (AE)
2. A characterization of serious adverse events (SAE)

Exploratory outcomes

1. Difference in VAS-pain at the 24-week follow-up visit between the intervention and placebo group.
2. Correlation between baseline quantitative sensory testing (QST) and treatment effect after 12 weeks.
3. Difference in QST change between the intervention and placebo group after 12 weeks of treatment.
4. Correlation between baseline psychosocial parameters, patient reported outcomes (PROMs) and treatment effect.
5. Difference in changes of the psychosocial parameters and PROMs between the intervention and control group after 12 weeks of treatment

Intervention: 10mg CBD tablets once daily for the first two weeks increasing to twice daily for week 3 and 4 if adequate analgesic effect is not attained at week 5 then the dose can be increased to 10mg thrice daily from week 5 and onward.

The medicine and placebo will be delivered and produced by Glostrup pharmacy.

Examination programme: All participants will receive a full medical interview and a physical examination which includes auscultation, blood pressure, heart rate and saturation measurements and BMI calculation. All participants will have blood drawn for later examination for markers of inflammation and degeneration. All participants will go through Quantitative Sensory Testing (QST). QST covers a wide range of different examinations techniques used to assess the functional status of the somatosensory system. In the present study pressure algometry and cuff algometry will be performed.

Pain phenotyping: Participants will answer a series of questionnaires related to the pain experience to assess: Anxiety and depression (the hospital anxiety and depression scale), pain catastrophizing (the pain catastrophizing scale), pain description (The short form McGill questionnaire and pain detect questionnaire), sleep quality (Pittsburgh sleep quality index) and a Widespread Pain Assessment questionnaire and the Symptom Severity Index. To assess function and quality of life the Short form 36 and Health assessment questionnaire will be used.

Patients with PsA: Will receive an examination for disease specific tests including: joint tenderness and swelling using the EULAR66/68 regiment, dactylitis evaluation using Leeds dactylitis index basic, skin involvement using the psoriasis area and severity index and nail psoriasis via nail psoriasis severity index.

Patients with Hand-OA: Will receive the following disease specific examinations evaluation of tender and swollen joints of the hands and wrists. Grip and pinch strength measurements using a hand-held dynamometer and the functional index of hand-osteoarthritis.

The trial consists of a screening visit, a baseline visit where the patient will undergo randomization, a phone consultation after 4 weeks a blood and urin sample after 6 weeks. and an end of trial visit at week 12. Patients will be invited to a follow-up visit at week 24.

Patients will be asked for adverse events at each visit and these are recorded in the eCRF.

ELIGIBILITY:
Inclusion Criteria Hand-OA:

* Patients (18 years or more) with Hand-OA according to the American Collage of Rheumatology (ACR) criteria (1990)
* Ability and willingness to give written informed consent and to meet the requirements of the study protocol.
* VAS pain during the last 24 hours 30mm or more
* Negative pregnancy test (serum HCG) prior to trial start (for women of childbearing potential) and the use of contraception throughout the study period and for 3 months after conclusion of the study period for males and females of childbearing potential. The forms of contraception include: intrauterine device (IUD) and hormonal contraceptives (contraceptive pill, implant, patch or injection or vaginal ring). Sterile and non-fertile participants do not have to use contraception. Sterile or non-fertile is defined as having undergone surgical sterilization (vasectomy / bilateral tubectomy, hysterectomy or bilateral oophorectomy) or post-menopausal status, defined as absence of menstrual period for at least 12 months prior to enrolment.

Inclusion criteria PsA

* Patients (18 years or more) with PsA according to the Calcification Criteria for Psoriatic Arthritis (CASPAR) criteria (2006)
* Ability and willingness to give written informed consent and to meet the requirements of the study protocol.
* VAS pain during the last 24 hours 30mm or more
* Negative pregnancy test (serum human chorionic gonadotropin (HCG)) prior to trial start and the use of contraception throughout the study period and for 1 month after conclusion of the study period for women of childbearing potential. The forms of contraception include: intrauterine device (IUD) and hormonal contraceptives (contraceptive pill, implant, patch or injection or vaginal ring). Sterile and non-fertile participants do not have to use contraception. Sterile or non-fertile is defined as having undergone surgical sterilization (vasectomy / bilateral tubectomy, hysterectomy or bilateral oophorectomy) or post-menopausal status, defined as absence of menstrual period for at least 12 months prior to enrolment.

Exclusion Criteria:

* Concurrent diagnosis of chronic regional pain syndrome or neuropathy
* Other known inflammatory rheumatic disease (i.e. rheumatoid arthritis, gout not in remission)
* Other known disease where exacerbations need to be treated with systemic corticosteroids (i.e. certain types of inflammatory bowel disease) or patients who have received systemic corticosteroid treatment during the last 3 months.
* Planning pregnancy, pregnant or breastfeeding. (Fertile women will be tested for pregnancy)
* Planned major surgery or recent major surgery (last 8weeks)
* Addictive behaviour or previously addictive behaviour defined as abuse of cannabis, opioids or other recreational or pharmaceutical drugs. Determined through patient interview and medical records.
* Contraindication to medical cannabis (Known allergy to ingredients, history of severe liver or kidney disease, history of schizophrenia or other serious psychiatric disease).
* Verified malignant disease
* History of epilepsy or severe cramps
* History of serious cardiovascular pathology
* Lacking ability to corporate with the research staff.
* Indication for changing the anti-inflammatory treatment regimen at baseline (PsA only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
VAS pain during the last 24 hours | Change from baseline to 12 weeks
  Measure with a 100mm Visual Analogue Scale (VAS) with higher values indicating more pain.

OTHER OUTCOMES:
Patients experiencing adverse events | 24 weeks
  Percentage of patients experiencing adverse events in placebo and intervention group
Characterization of serious adverse events | 24 weeks
  Description of which serious adverse events where experience in each group
Difference in VAS-pain at the 24-week follow-up visit between the intervention and placebo group. | at 24week followup
  Measure with a 100mm Visual Analogue Scale (VAS) with higher values indicating more pain.
Correlation between baseline quantitative sensory testing (QST) and treatment effect after 12 weeks. | at 12week visit
  QST measurements will include pain detection threshold, pain tolerance threshold, temporal summation and conditioned pain modulation
Correlation between baseline psychosocial parameters, patient reported outcomes (PROMs) and treatment effect | at 12 week visit
  patient reported outcome includes: Expected effect of treatment is measured using the Stanford expectations scale. Pain catastrophizing thoughts are measured using the Pain catastrophizing scale. Presence of widespread pain is evaluated using the Widespread Pain Index and the Symptom Severity Scale. Sleep quality is evaluated using the Pittsburgh Sleep Quality Index. Presence of anxiety and depression is measured using the Hospital Anxiety and Depression Scale. Furthermore, pain phenotype will be quantified using the Pain Detect Questionnaire and Short Form McGill questionnaire. Quality of life is quantified using the Short form 36 and disability using the Health Assessment Questionnaire Disability Index and Functional index of hand osteoarthritis.
5. Difference in changes of the psychosocial parameters and PROMs between the intervention and control group after 12 weeks of treatment | at 12 week visit
  patient reported outcome includes: Expected effect of treatment is measured using the Stanford expectations scale. Pain catastrophizing thoughts are measured using the Pain catastrophizing scale. Presence of widespread pain is evaluated using the Widespread Pain Index and the Symptom Severity Scale. Sleep quality is evaluated using the Pittsburgh Sleep Quality Index. Presence of anxiety and depression is measured using the Hospital Anxiety and Depression Scale. Furthermore, pain phenotype will be quantified using the Pain Detect Questionnaire and Short Form McGill questionnaire. Quality of life is quantified using the Short form 36 and disability using the Health Assessment Questionnaire Disability Index and Functional index of hand osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Vela, Principal Investigator — Dept. of rheumatology Aalborg University Hospital
Locations (1):
- Department of Rheumatology Aalborg Universityhospital North, Aalborg, Denmark